CLINICAL TRIAL: NCT02471755
Title: A Randomized Pilot Study of Electro-acupuncture for Menopausal Transition Symptoms
Brief Title: Electro-acupuncture for Menopausal Transition Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, xiaoxuliu, doctor, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012BAI24B01-012
Record Dates: First submitted 2015-06-07; First posted 2015-06-15 (Estimated); Results first posted 2015-11-23 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-10

CONDITIONS: Menopause
Keywords: electro-acupuncture; menopause; menopausal transition symptoms; efficacy; RCT; placebo control

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electro-acupuncture Group (Active Comparator)
  Interventions: Device: Eelectro-acupuncture
- Sham Electro-acupuncture Group (Placebo Comparator)
  Interventions: Device: Sham Eelectro-acupuncture

INTERVENTIONS:
Device: Eelectro-acupuncture — The bilateral acupoints of EX-CA1, ST25, SP6 and RN4 were selected for the treatment program.After regular disinfection,adhesive pads were placed on surface of all these acupoints. For RN4, EX-CA1, ST25, needles (0.30*75mm) were inserted into the points vertically throughout the pads, skin, fat tissue, and abdominal muscles until the participant had feeling of pricking. For SP6, needles were inserted into the acupoint to a depth of 1 cun,accompanied by manipulation of lifting, thrusting, and twisting 3 times. Electronic stimulator was connected to EX-CA1 and ST25 with dilatational wave, 10/50HZ, 0.1 to 1.0mA. The current intensity was adjusted to abdomen shivering without pain. Treatment lasted for 30 minutes and acupuncture manipulation for RN4 and SP6 were performed every 10 minutes.
  Arms: Electro-acupuncture Group
Device: Sham Eelectro-acupuncture — Non-acupoints approximate to RN4, ST25, EX-CA1 and SP6 were selected bilaterally, and adhesive pads were placed on the surface of selected non-acupoints' location. Blunt needles were inserted into the pads and to touch, rather than penetrate the surface of skin. Meanwhile, like EA group, manipulations of lifting, thrusting and twisting on non-acupoint approximate to RN4 and SP6 were performed 3 times. Sham Electronic stimulator was applied to the non-acupoint approximate to EX-CA1 and ST25, providing the outward appearance of the procedure in EA group but with no current intensity actually applied. Any other interventions were rigorously maintained the same as in the EA group.
  Arms: Sham Electro-acupuncture Group

SUMMARY:
This trial aimed at exploring the efficacy as well as safety of electro-acupuncture for MT symptoms.

DETAILED DESCRIPTION:
This was a RCT pilot study to assess the efficacy of Electro-acupuncture for menopausal transition participants.90 patients were randomly assigned to electro-acupuncture or sham electro-acupuncture group with a ratio of 1:1.During the whole process,all participants, evaluators and statisticians apart from acupuncturists remained strictly blinded.The changes of average 24 h hot flash scores of week8 from baseline was set as primary outcome. With statistical power of 90%, and a two-sided α at 0.05, as well as a drop-out rate less than 20%, sample size was estimated at 90 participants. Data analysis was based on ITT principles, and 89 participants were included in data analysis(1 participant didn't want to participate).According to methods of LOCF, missing data were imputed to fill any gaps according to the last visit. For comparison between baseline and treatment (average 24h hot flash scores, MRS, hormone levels), data was tested by the t test or nonparametric test; for comparison between two independent samples, data were tested with t test, nonparametric test or X2 test. P<0.05 was regarded as statistically significance.

ELIGIBILITY:
Inclusion Criteria:

* Participants meeting the following criteria were included in study:

  1. Had a diagnosis of MT (cycle length irregularity: 7 days earlier or later than usual, the last menstruation was no longer than 11 month earliar over the previous year; Specific symptoms of MT: hot flashes, night sweating, insomnia, sexual problems, anxiety, depression etc.);
  2. Aged from 40 to 55 years old;
  3. Pregnancy test was negative;
  4. Participants were informed about the study and signed a consent form voluntarily.

     Exclusion Criteria:
* Participants with any of the following criteria were omitted from the study:

  1. 3 month regular cycle length before enrollment;
  2. Took drugs for treatment in past month like estrogen, soybeans isoflavone, SSRIs, progestin, black sesame or vitamin E;
  3. Ovarian and uterine disease: ovarian cyst, uterine myoma more than 4cm in diameter, history of ovariectomy or hysterectomy;
  4. Willing or plan to become pregnant or to breast-feed;
  5. Regular took sedatives or anxiolytics;
  6. Habitual smoker or heavy alcoholic;
  7. Severe disease: history of radio-chemotherapy, coagulation disorders, severe dysfunction of liver or kidney, application of cardiac pacemaker or artificial joints, insufficiency controlled hypertension, diabetes, thyroid diseases, malignant tumor and psychiatric problems).

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, Doctor, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This prospective RCT was conducted at Guang'anmen Hospital, China Academy of Chinese Medical Sciences (Beijing, China), from April 2013 to December 2014. Participants with MT were recruited via hospital posters.
Pre-assignment Details: A total of 192 participants were assessed for eligibility; 102 participants were excluded from the trial(53 didn't meet inclusion criteria, 26 declined to participate the trial, 23 for other reasons). 90 participants were randomly allocated to the EA group or the sham EA group.
Period: Overall Study
Arm/Group | Electro-acupuncture Group | Sham Electro-acupuncture Group
Started | 45 | 45
Completed | 44 | 44
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Electro-acupuncture Group | Sham Electro-acupuncture Group | Total
Number analyzed (Participants) | 44 | 45 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.05 (4.41) | 50.69 (3.79) | 50.84 (4.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 45 | 89
  Male | 0 | 0 | 0
Educational Level [Number; unit: participants]
  Preliminary education | 0 | 1 | 1
  Secondary education | 33 | 25 | 58
  Tertiary education | 11 | 19 | 30
Weight [Mean (Standard Deviation); unit: Kg] | 58.02 (5.66) | 57.66 (7.95) | 57.84 (6.87)
Height [Mean (Standard Deviation); unit: cm] | 159.39 (3.87) | 159.49 (3.88) | 159.44 (3.85)
Menopausal Course [Median (Inter-Quartile Range); unit: month] | 16.00 [12.00 to 18.00] | 16.00 [12.50 to 24.00] | 16.00 [12.00 to 21.00]
Menopausal Stage [Number; unit: participants] — According to different cycle lengths, MT can be divided into two stages: early MT (>7 days different from normal) and late MT (≥60 days, 2 skipped cycles, 1 interval of amenorrhea).
  participants
    Early stage | 17 | 24 | 41
    Late stage | 27 | 21 | 48
Ever Received Drug Therapy [Number; unit: participants]
  Yes | 5 | 1 | 6
  No | 39 | 44 | 83
24 h Hot Flash Score [Median (Inter-Quartile Range); unit: Scores on a scale] — Hot flash scores are calculated as (hot flash frequency x severity)/7, with severity scores ranging from 1=mild 2=moderate to 3=severe.
  Scores on a scale | 8.07 [4.78 to 12.50] | 7.26 [5.31 to 11.93] | 7.71 [5.15 to 12.22]
Menopause Rating Scale [Median (Inter-Quartile Range); unit: Scores on a scale] — The MRS is composed of 11 items to assess menopausal symptoms, and each item is graded from 0 (no symptoms) to 4 (very severe symptoms). As a result, the scores of the MRS range from 0 to 44, with higher scores indicating more severe symptoms.
  Scores on a scale | 17.50 [12.25 to 19.75] | 15.00 [11.00 to 19.50] | 16.00 [11.50 to 19.50]
FSH [Median (Inter-Quartile Range); unit: mIU/ml] | 42.85 [31.16 to 51.96] | 44.47 [36.13 to 48.59] | 44.12 [35.72 to 49.28]
LH [Median (Inter-Quartile Range); unit: mIU/ml] | 33.08 [20.92 to 43.21] | 32.89 [22.26 to 37.50] | 32.89 [21.34 to 38.75]
FSH/LH [Median (Inter-Quartile Range); unit: ratio] | 1.38 [0.90 to 1.67] | 1.44 [1.11 to 1.69] | 1.42 [0.99 to 1.67]
E2 [Median (Inter-Quartile Range); unit: pmol/l] | 73.73 [42.03 to 110.54] | 51.38 [37.56 to 92.18] | 65.77 [38.57 to 103.39]

OUTCOME MEASURES:

1. Primary Outcome: Change of Average 24 h Hot Flash Score From Baseline
Description: Every day during the 4th, 8th, 20th, and 32nd weeks, symptoms and specific times of hot flashes were recorded in hot flash diaries by the participants.Data from weeks 4, 20 and 32 were recorded as the second time frame.According to the severity categories suggested by Food and Drug Administration (FDA), hot flashes were assessed as mild, moderate, or severe. Hot flash scores are calculated as (hot flash frequency x severity)/7, with severity scores ranging from 1=mild 2=moderate to 3=severe.
Time Frame: week8;wee4,20,32
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Electro-acupuncture Group | Sham Electro-acupuncture Group
Number analyzed (Participants) | 44 | 45
Scores on a scale
  week8 | -2.29 [-4.79 to -0.47] | -0.71 [-3.28 to 0.09]
  week4 | -0.78 [-2.54 to 0.00] | -0.71 [-2.72 to 0.34]
  week20 | -2.43 [-4.90 to -0.86] | -1.14 [-4.00 to 0.50]
  week32 | -3.79 [-6.00 to -1.14] | -0.87 [-4.57 to 0.14]

2. Secondary Outcome: Change of MRS (Menopause Rating Scale) From Baseline
Description: MRS(Menopause Rating Scale) was designed to measure MT symptoms and to explore the influences on life qualities in a standardized way. In MRS, symptoms such as impaired memory, depression, insomnia, sweating, hot flashes, nervousness, joints complaints, lack of concentration were evaluated and calculated in numbers to describe the situation of patient. Scores on MRS range from 0 to 44, with higher scores indicating more severe symptoms.
Time Frame: week8;wee4,20,32
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Electro-acupuncture Group | Sham Electro-acupuncture Group
Number analyzed (Participants) | 44 | 45
Scores on a scale
  week8 | -4.00 [-9.00 to -1.25] | -6.00 [-9.00 to 0.00]
  week4 | -1.50 [-5.75 to 0.75] | -4.00 [-6.50 to 0.00]
  week20 | -6.00 [-11.00 to -1.00] | -5.00 [-8.50 to -1.00]
  week32 | -7.00 [-12.75 to -2.00] | -5.00 [-10.00 to -0.50]

3. Secondary Outcome: Change of FSH From Baseline
Description: Serum sample of participants was examined at the 2nd to 4th day of menstrual period; if the participant was not in menstrual period, Serum sample would be tested in coming cycle length; for participants in menopause period, Serum sample was examined at the end of the week of 8th and 20th.
Time Frame: week8,week20
Measure: Median (Inter-Quartile Range); unit: mIU/ml
Arm/Group | Electro-acupuncture Group | Sham Electro-acupuncture Group
Number analyzed (Participants) | 44 | 45
mIU/ml
  week8 | -1.90 [-9.98 to 10.03] | 0.70 [-1.87 to 11.04]
  week20 | -1.69 [-11.11 to 24.22] | 1.93 [-0.58 to 18.67]

4. Secondary Outcome: Change of LH From Baseline
Description: as for outcome 3
Time Frame: week8,week20
Measure: Median (Inter-Quartile Range); unit: mIU/ml
Arm/Group | Electro-acupuncture Group | Sham Electro-acupuncture Group
Number analyzed (Participants) | 44 | 45
mIU/ml
  week8 | -2.58 [-7.99 to 3.61] | 0.99 [-3.01 to 4.78]
  week20 | -0.66 [-8.56 to 11.11] | 0.79 [-0.13 to 9.74]

5. Secondary Outcome: Change of FSH/LH From Baseline
Description: as for outcome 3
Time Frame: week8,week20
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Electro-acupuncture Group | Sham Electro-acupuncture Group
Number analyzed (Participants) | 44 | 45
ratio
  week8 | 0.10 [-0.10 to 0.33] | -0.01 [-0.15 to 0.24]
  week20 | 0.06 [-0.20 to 0.33] | -0.01 [-0.10 to 0.18]

6. Secondary Outcome: Change of E2 From Baseline
Description: as for outcome 3
Time Frame: week8,week20
Measure: Median (Inter-Quartile Range); unit: pmol/l
Arm/Group | Electro-acupuncture Group | Sham Electro-acupuncture Group
Number analyzed (Participants) | 44 | 45
pmol/l
  week8 | 2.92 [0.00 to 28.37] | 0.40 [-1.88 to 12.16]
  week20 | 13.75 [-1.22 to 62.76] | 2.43 [-14.56 to 31.38]

ADVERSE EVENTS:
Time Frame: 32 weeks
Arm/Group | Electro-acupuncture Group | Sham Electro-acupuncture Group
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/45
Other Adverse Events (participants affected / at risk) | 3/44 | 2/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Electro-acupuncture Group (N=44) | Sham Electro-acupuncture Group (N=45)
Headache (Nervous system disorders) | 1 | 1
sore throat (General disorders) | 1 | 0
arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
fatigue (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No